CLINICAL TRIAL: NCT00695396
Title: A Randomized, Double Blind, Placebo Controlled, Multicenter Study Evaluating Epoetin Alfa Initiated at 40,000 IU Every Week or 80,000 IU Every Week Versus Placebo in Subjects With IPSS Low- or Intermediate-1 Risk Myelodysplastic Syndromes at Risk For Transfusion
Brief Title: A Study Evaluating Epoetin Alfa 40,000 IU (International Units) Every Week or 80,000 IU Every Week Compared to Placebo in Patients With Low or Intermediate-1 Risk Myelodysplastic Syndromes at Risk for Transfusion
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped due to low subject enrollment. No safety issue or other concern factored into this decision.
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Centocor Ortho Biotech Services, L.L.C. (Industry)
Responsible Party: CDTL PROCURIT/EPREX, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR013651; EPOANE3018
Record Dates: First submitted 2008-06-05; First posted 2008-06-11 (Estimated); Results first posted 2011-03-17 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Myelodysplastic Syndromes; Anemia
Keywords: MDS; Myelodysplastic syndromes; Anemia; Epoetin alfa; EPO
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 001 (Experimental): Epoetin alfa 40 000 IU subcutaneously once every week (1 mL dose) for 48 weeks
  Interventions: Drug: Epoetin alfa
- 002 (Experimental): Epoetin alfa 80 000 IU subcutaneously once every week (2 mL dose) for 48 weeks
  Interventions: Drug: Epoetin alfa
- 003 (Placebo Comparator): Placebo Matching volume 1 mL for 48 weeks
  Interventions: Drug: Placebo
- 004 (Placebo Comparator): Placebo Matching volume 2 mLfor 48 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Matching volume 2 mLfor 48 weeks
  Arms: 004
Drug: Epoetin alfa — 40,000 IU subcutaneously once every week (1 mL dose) for 48 weeks
  Arms: 001
Drug: Placebo — Matching volume 1 mL for 48 weeks
  Arms: 003
Drug: Epoetin alfa — 80,000 IU subcutaneously once every week (2 mL dose) for 48 weeks
  Arms: 002

SUMMARY:
The purpose of this study is to demonstrate that Epoetin alfa treatment reduces red blood cell transfusions in anemic patients with myelodysplastic syndromes (MDS). Myelodysplastic syndromes are a group of disorders characterized by progressive bone marrow failure and an increased risk of development of leukemia.

DETAILED DESCRIPTION:
This is a randomized (patients are assigned by chance to a treatment group), double-blind (neither the patient or the physician know which treatment is being received by the patient), placebo-controlled, multicenter study of epoetin alfa in anemic patients who are diagnosed with myelodysplastic syndromes (MDS) according to protocol-specified criteria. Patients meeting entry criteria for the study will be randomly assigned to receive epoetin alfa 40,000 IU or 80,000 IU or a matching volume of placebo administered by subcutaneous (under the skin) injection once every week. Doses of study drug will be withheld, decreased, or increased on the basis of weekly hemoglobin concentrations monitored in patients and predefined dose adjustment guidelines. An Independent Data Monitoring Committee (IDMC) will periodically review study data and for the assessment of disease progression, an independent central reviewer will review bone marrow specimens and peripheral blood counts. Safety will be monitored throughout the study at predetermined intervals and as clinically indicated by physical examination, laboratory tests and evaluation of adverse events. Patients in the Treatment Phase will be randomly assigned to receive once weekly epoetin alfa subcutaneously (SC) at a dose of 40,000 IU (1 mL) or 80,000 IU (2ML) or matching volume of placebo (1 mL or 2 mL) once every week for 48 weeks. Patients may continue to receive double-blinded treatment after 48-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS according to protocol-specified criteria via bone marrow studies performed within 12 weeks before randomization

Exclusion Criteria:

* No prior or concurrent treatment with epoetin alfa or any other approved or experimental erythropoietin stimulating agents (ESAs) within the previous 12 months before randomization
* No prior use of approved or experimental agents for the treatment of MDS or recent treatment with granulocyte colony stimulating factor (G-CSF) or granulocyte macrophage colony stimulating factor (GM-CSF) for the treatment of neutropenia
* Patients must not have secondary MDS or anemia caused by factors other than MDS (including iron deficiency, vitamin B12 or folate deficiencies, hemolysis, chronic renal failure, or gastrointestinal bleeding)
* No history (within 12 months) of deep venous thrombosis
* or history (within 6 months) of stroke, acute coronary syndrome or other arterial thrombosis
* Not currently receiving therapeutic anticoagulants or have uncontrolled hypertension
* No uncontrolled disease or dysfunction deemed clinically significant by the Investigator not attributable to MDS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: (1ml or 2 mL) subcutaneously once every week
- Epoetin Alfa 40000 IU: (1 mL) subcutaneously once every week
- Epoetin Alfa 80000 IU: (2 mL) subcutaneously once every week
Period: Overall Study
Arm/Group | Placebo | Epoetin Alfa 40000 IU | Epoetin Alfa 80000 IU
Started | 8 | 8 | 9
Completed | 1 | 0 | 1
Not Completed | 7 | 8 | 8
Not completed — Study Closed Prematurely | 5 | 6 | 8
Not completed — Withdrawal by Subject | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Epoetin Alfa 40000 IU | Epoetin Alfa 80000 IU | Total
Number analyzed (Participants) | 8 | 8 | 9 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 4
  >=65 years | 7 | 7 | 7 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 73 (10.52) | 77.3 (9.78) | 67.7 (9.89) | 72.4 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 7 | 12
  Male | 6 | 5 | 2 | 13
Region of Enrollment [Number; unit: participants]
  CANADA | 1 | 0 | 0 | 1
  ITALY | 0 | 1 | 0 | 1
  RUSSIA | 2 | 0 | 4 | 6
  USA | 5 | 7 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Red Blood Cell (RBC) Transfusion
Description: Incidence of participants who received at least 1 Red Blood Cell (RBC) transfusion during the study (from randomization through the end of study)
Time Frame: Approximately 48 weeks
Population: The intent-to-treat (ITT) population was defined as all participants randomly assigned to a treatment group, regardless of whether they received any treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | Epoetin Alfa 40000 IU | Epoetin Alfa 80000 IU
Number analyzed (Participants) | 8 | 8 | 9
participants | 5 | 3 | 1

2. Secondary Outcome: RBC Transfusion From Day 29 Through the End of Study
Description: incidence of participants who received at least 1 RBC transfusion from Day 29 through the end of study (approximately 48 weeks).
Time Frame: Day 29 through the end of study (approximately 48 weeks)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Epoetin Alfa 40000 IU | Epoetin Alfa 80000 IU
Number analyzed (Participants) | 8 | 8 | 9
participants | 4 | 2 | 1

3. Secondary Outcome: Transfusion Dependent
Description: Participants who were transfusion-dependent were those who received 4 or more RBC units during a consecutive 8-week period.
Time Frame: Approximately 48 weeks
Population: The intent-to-treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | Placebo | Epoetin Alfa 40000 IU | Epoetin Alfa 80000 IU
Number analyzed (Participants) | 8 | 8 | 9
participants | 2 | 2 | 1

ADVERSE EVENTS:
Arm/Group | Placebo | Epoetin Alfa 40000 IU | Epoetin Alfa 80000 IU
Serious Adverse Events (participants affected / at risk) | 2/8 | 2/8 | 4/9
Other Adverse Events (participants affected / at risk) | 7/8 | 4/8 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | Epoetin Alfa 40000 IU (N=8) | Epoetin Alfa 80000 IU (N=9)
Aplasia Pure Red Cell (Blood and lymphatic system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | Epoetin Alfa 40000 IU (N=8) | Epoetin Alfa 80000 IU (N=9)
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Oral Pain (Gastrointestinal disorders) | 1 | 0 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 2 | 1
Asthenia (General disorders) | 1 | 0 | 2
Hyperthermia (General disorders) | 0 | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 1
Blood Urine Present (Investigations) | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Because this study was terminated prematurely due to slow enrollment, only limited data were collected. No formal statistical testing was performed. Only descriptive statistics were provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No